CLINICAL TRIAL: NCT00000828
Title: Study of Perinatal Transmission of Zidovudine-Resistant HIV Among Pregnant Women Treated With Zidovudine
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 255
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Pregnancy Complications, Infectious; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Drug Resistance, Microbial; Disease Transmission, Vertical
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious; Acquired Immunodeficiency Syndrome; AIDS-Related Complex

SUMMARY:
To identify patterns of zidovudine ( AZT ) susceptibility among mother/infant pairs with perinatal HIV transmission.

Most HIV-infected infants acquire their disease via perinatal transmission. Since transmission of HIV-resistant strains to infants could alter the course of disease and response to currently recommended treatment, a study to assess the patterns of AZT susceptibility among mother/infant pairs with perinatal transmission is essential to delineate future therapeutic strategies.

DETAILED DESCRIPTION:
Most HIV-infected infants acquire their disease via perinatal transmission. Since transmission of HIV-resistant strains to infants could alter the course of disease and response to currently recommended treatment, a study to assess the patterns of AZT susceptibility among mother/infant pairs with perinatal transmission is essential to delineate future therapeutic strategies.

HIV-infected pregnant women are enrolled at 20-36 weeks gestation. Patients have blood drawn for HIV culture at study entry and at delivery. Infants have blood drawn for HIV culture at delivery and at 1, 3, 6, and 18 months of age.

ELIGIBILITY:
Inclusion Criteria

Prior Medication: Required:

* At least 6 months of prior AZT, including continuously during the current pregnancy.

Patients must have:

* HIV seropositivity.
* CD4 count <= 300 cells/mm3.
* Gestational age of 20-36 weeks, with intention to carry pregnancy to term.
* At least 6 months of prior AZT therapy, including continuous AZT therapy during the current pregnancy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Evidence of pre-existing fetal anomalies that would preclude survival to the end of the study, such as anencephaly, renal agenesis, or Potter's syndrome.

Concurrent Medication:

Excluded:

* Antiretrovirals other than AZT.

Ages: 13 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250

CONTACTS AND LOCATIONS:
Overall Officials: Bardeguez AD, Study Chair; Pitt J, Study Chair
Locations (29):
- United States (28):
  - Univ of Alabama at Birmingham Schl of Med / Pediatrics, Birmingham, Alabama
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Connecticut Children's Med Ctr - Pediatric, Hartford, Connecticut
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Miami (Pediatric), Miami, Florida
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ Hosp, New Orleans, Louisiana
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Columbus Children's Hosp, Columbus, Ohio
- San Juan City Hosp, San Juan, Puerto Rico

REFERENCES:
- [Background] Bardeguez AD. Management of HIV infection for the childbearing age woman. Clin Obstet Gynecol. 1996 Jun;39(2):344-60. doi: 10.1097/00003081-199606000-00009. No abstract available. PMID 8734001
- [Background] Bardeguez AD, Taylor U, Appuzio J, Leus C, Lister M, Denny T, Palumbo P, Connor E. Characteristics of pregnant women infected with human immunodeficiency virus 1: Newark perinatal transmission study. Int Conf AIDS. 1991 Jun 16-21;7(2):193 (abstract no WB2044)
- [Background] Japour AJ, Welles S, McIntosh K, Colson A, Chung P, Lockman S, Davenny K, Fowler MG, Hansen IC, Kalish L, Moye J, Rick K, Zorilla C, Pitt J. ZDV resistance (ZDVR) mutations in ZDV exposed mother infant pairs: preliminary findings from the women and infants transmission study (WITS). Int Conf AIDS. 1996 Jul 7-12;11(1):370 (abstract no TuC2606)
- [Background] Garcia PM, Kalish LA, Pitt J, Minkoff H, Quinn TC, Burchett SK, Kornegay J, Jackson B, Moye J, Hanson C, Zorrilla C, Lew JF. Maternal levels of plasma human immunodeficiency virus type 1 RNA and the risk of perinatal transmission. Women and Infants Transmission Study Group. N Engl J Med. 1999 Aug 5;341(6):394-402. doi: 10.1056/NEJM199908053410602. PMID 10432324